CLINICAL TRIAL: NCT05491746
Title: Diabetic Retinopathy Tethered Augmented Reality With Eye4 Study
Acronym: DRTARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyedaptic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Retinopathy; Low Vision
MeSH Terms: conditions — Diabetic Retinopathy; Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye4 (Experimental): This is the arm with the Eyedaptic Device
  Interventions: Device: Eye4
- Baseline (Placebo Comparator): This is the placebo arm with the best correction the subject has
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Eye4 — Patients will see if the device helps them see better at distance and near and if it improves their contrast sensitivity.
  Arms: Eye4
Other: Placebo — This is the patient's best corrected vision with or without glasses/contact lenses
  Arms: Baseline

SUMMARY:
Diabetes has reached epidemic levels in North America and with it, diabetic retinopathy is increasingly affecting the vision of millions of people. Despite treatment many patients still have vision loss that cannot be improved medically or with prescription eyeglasses. Our study is going to look at an FDA Class 1 Exempted visual aid that uses augmented reality to help people see better.

DETAILED DESCRIPTION:
In this study subjects will have their best corrected visual acuity and contrast sensitivity compared to their best vision and contrast with the Eyedaptic device. The Eyedaptic device is an FDA 510(k) Class 1 Exempt device as it is a visual aid. This is a pilot study to determine whether subjects with diabetic retinopathy associated vision loss obtain a benefit with augmented reality vision.

Subjects will receive a manifest refraction. When subjects have their optimal corrective lenses, the subjects' vision will be tested with their corrective lenses alone and again using the Eyedaptic device. This will be a single visit study, with no follow up.

ELIGIBILITY:
Inclusion Criteria:

* Best correct visual acuity in the better seeing eye between 20/60 and 20/800
* History of diabetic retinopathy

Exclusion Criteria:

* Unable to complete the visit
* Unable to give a reliable measurement of vision
* Unable to comfortably wear the glasses for at least 60 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity at distance | Day 1
  Visual acuity at distance using Snellen Visual Acuity Chart

SECONDARY OUTCOMES:
Visual acuity at near | Day 1
  Visual acuity at near tested using Ridgevue Near Vision chart
Contrast sensitivity | Day 1
  Contrast sensitivity measured using the Ridgevue contrast sensitivity scale

CONTACTS AND LOCATIONS:
Overall Officials: Mitul Mehta, MD, Principal Investigator — Eyedaptic
Locations (1):
- Eyedaptic, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No